CLINICAL TRIAL: NCT00973765
Title: Randomized Placebo-Controlled Trial of Bactrim on 7 Day Outcome in Emergency Department Patients With Uncomplicated Abscesses at Risk for Community Acquired Methicillin Resistant Staph Aureus
Brief Title: Prospective Randomized Trial of Bactrim on 7 Day Outcome in Patients With Uncomplicated Abscesses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Gillian Schmitz, MD, Wilford Hall Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWH20080055H_
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Results first posted 2010-03-02 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2009-09

CONDITIONS: Abscesses
Keywords: abcess; MRSA; cellulitis; antibiotics; uncomplicated abscesses
MeSH Terms: conditions — Abscess; Cellulitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bactrim DS (800/160) 2 pills po BID x 7 days (Active Comparator): active comparator
  Interventions: Drug: bactrim
- Matched placebo 2 pills po BID x 7 days (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bactrim — bactrim DS (800/160) 2 pills PO BID x 7 days
  Arms: bactrim DS (800/160) 2 pills po BID x 7 days
Drug: placebo — placebo 2 pills po BID x 7 days
  Arms: Matched placebo 2 pills po BID x 7 days

SUMMARY:
Patients will be enrolled in a multi-center study to prospectively evaluate outcome after treatment for an uncomplicated skin abscess. All patients will receive incision and drainage and wound cultures. Patients will then be randomized to 1) placebo two tablets PO BID X 7 days or 2) bactrim DS (800/160) two tablets PO BID x 7 days. Patients will then return to the emergency department ED) at 48 hours and 7 for wound repacking and evaluation. The primary outcome is treatment failure rates at 7 days after incision and drainage. Patients who are clinically worsening or not improving after 48 hours will then be treated with additional antibiotics or admission if needed. Data will be analyzed both by initial randomization and intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include all patients age 16 and older who present to the emergency department with a skin abscess that requires incision and drainage.

Exclusion Criteria:

* Exclusion criteria include patients with diabetes, HIV, cancer or other immunocompromised patients.
* Additionally, any patients who received antibiotics within one week of presentation or were hospitalized in previous month will be excluded to minimize potential confounding variables.
* Pregnant and breastfeeding patients will also be excluded due to possible safety concerns with antibiotic treatment.
* Patients with abscesses on face, perirectal, or perianal regions, abscesses with known tracks or fistulas to deeper structures, or abscesses requiring surgical drainage in an operating room are excluded.
* Patients with fever or evidence of systemic infection
* Finally, patients with sulfa allergy will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilford Hall Medical Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Derived] Schmitz GR, Bruner D, Pitotti R, Olderog C, Livengood T, Williams J, Huebner K, Lightfoot J, Ritz B, Bates C, Schmitz M, Mete M, Deye G. Randomized controlled trial of trimethoprim-sulfamethoxazole for uncomplicated skin abscesses in patients at risk for community-associated methicillin-resistant Staphylococcus aureus infection. Ann Emerg Med. 2010 Sep;56(3):283-7. doi: 10.1016/j.annemergmed.2010.03.002. Epub 2010 Mar 26. PMID 20346539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 1, 2008 - June 1, 2009 in emergency department
Groups:
- Active Comparator: Bactrim DS (800/160) 2 pills po BID x 7 days
- Placebo: Matched placebo 2 pills po BID x 7 days
Period: Overall Study
Arm/Group | Active Comparator | Placebo
Started | 96 (96) | 116 (116)
Completed | 88 (88) | 102 (102)
Not Completed | 8 | 14
Not completed — Lost to Follow-up | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Placebo | Total
Number analyzed (Participants) | 96 | 116 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 94 | 116 | 210
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 31.5 (13.3) | 31.1 (12.5) | 31.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 44 | 72
  Male | 68 | 72 | 140
Region of Enrollment [Number; unit: participants]
  United States | 96 | 116 | 212

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failures at 7 Days
Description: worsening abscess or new recurrence of abscess
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Active Comparator | Placebo
Number analyzed (Participants) | 96 | 116
participants | 15 | 27

ADVERSE EVENTS:
Arm/Group | Active Comparator | Placebo
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/212
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No